CLINICAL TRIAL: NCT06045598
Title: Investigation of the Influence of Postural Control, Ankle and Trunk Proprioception in Patients With Type 2 Diabetes
Brief Title: Postural Control, Ankle and Trunk Proprioception in Type 2 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Günseli Usgu, Principal Investigator, Hasan Kalyoncu University
Other Study IDs: HKU 2023
Record Dates: First submitted 2023-08-23; First posted 2023-09-21 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Type2diabetes
Keywords: type 2 diabetes; postural control; proprioception; sensation; cognition
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- type 2 diabetes group: Participants between the ages of 18-65 who have been diagnosed with Type 2 diabetes according to the criteria of the American Diabetes Association (ADA).
  Interventions: Other: Semmes Weinstein Monofilament Test; Other: Proprioception measurement; Other: Postural control assessment; Other: Dynamic balance assessment; Other: Timed Up and Go Test; Other: Montreal Cognitive Assessment
- control group: Healthy participants between the ages of 18-65 who have not been diagnosed with Type 2 diabetes
  Interventions: Other: Semmes Weinstein Monofilament Test; Other: Proprioception measurement; Other: Postural control assessment; Other: Dynamic balance assessment; Other: Timed Up and Go Test; Other: Montreal Cognitive Assessment

INTERVENTIONS:
Other: Semmes Weinstein Monofilament Test — The 10 g Semmes-Weinstein monofilament assessment (SWME) is used to assess sensory loss and screen for diabetic neuropathy. In our study, the evaluation will be made on the plantar surfaces of the 1st fingers, the plantar surfaces of the 1st, 3rd, and 5th metatarsal heads, and the plantar surfaces of the heel in the right and left feet. The first force value felt will be taken as the evaluation data.
Other: Proprioception measurement — Ankle proprioception will be measured with the participant's knees lying on their back in a semi-flexed position. The test will be performed for 10 degrees of dorsiflexion and 20 degrees of plantar flexion, respectively. Measurements will be made with an electrogoniometer device. The difference between the required degree and the degree in the position brought by the participant will be taken as evaluation data.
  Lumbal region proprioception measurement will be made with lumbar flexion and extension movements. The participant will be asked to perform active lumbar flexion. Then, lumbar flexion movement will be performed up to 50% of the measured active flexion angle and it will be requested to stay in this position for 10 seconds. After the participant returns to the upright position, he will be asked to come back to the learned angle and the difference in angle will be taken as evaluation data. The same procedure will be done for the lumbar extension movement.
Other: Postural control assessment — Postural control evaluation will be done with the Gyko-Microgate software. Bluetooth data transmission enables real-time measurements to be transferred directly to the computer. After the device was placed on the body of the person thanks to the wearable vest, a connection was established with the software on the computer.
  To evaluate postural control, with eyes open, eyes closed and eyes open on a hard surface, accompanied by a cognitive dual task; On soft ground, with eyes open, eyes closed and eyes open, the person is asked to remain in a stable balance for 30 seconds, accompanied by a cognitive dual task. For the cognitive dual task, two countdowns and K-A-S verbal fluency exercises will be performed in each assessment. As a result of each evaluation, data on ellipsoid area, anteroposterior velocity, anteroposterior distance, mediolateral velocity, and mediolateral distance will be obtained.
Other: Dynamic balance assessment — Dynamic balance evaluation will be done with the Gyko device. To evaluate dynamic balance, walking with eyes open on hard ground, walking with cognitive dual task on hard ground; walking with eyes open on soft ground, and cognitive dual task on soft ground will be evaluated. The walking distance is determined as 6 meters. The first 1 meter and the last 1 meter will not be taken into consideration. The measurement will start at the 1st meter and end at the 5th meter. The measurement will be carried out at a distance of 4 meters. As a cognitive task, the participants will be given the task of counting down by two and K-A-S verbal fluency. As a result of each evaluation, data on the ellipsoid area, anteroposterior velocity, anteroposterior distance, mediolateral velocity, and mediolateral distance will be obtained.
Other: Timed Up and Go Test — The Timed Get Up and Walk Test is used to assess balance and fall risk. The participant stands up from the chair, walks 3 meters, turns back, and sits back on the chair. The time elapsed during these phases was recorded.
  In our study, the patient will be asked to start the test after the Gyko device is fixed with a wearable vest. During the test, data on the ellipsoid area, anteroposterior velocity, anteroposterior distance, mediolateral velocity, and mediolateral distance will be taken.
Other: Montreal Cognitive Assessment — MoCA is a 10-minute scale that measures global cognitive skills. It includes items consisting of attention and concentration, executive functions, memory, language, visuospatial skills, abstract thinking, calculation and orientation skills. The lowest score that can be obtained from the scale is 0, and the highest score is 30. Scores of 21 and below indicate the presence of cognitive impairment.

SUMMARY:
The investigators aim to assess the postural control, ankle, and trunk proprioception, plantar sensation, and general cognitive status in patients with Type 2 diabetes.

DETAILED DESCRIPTION:
The investigators aim to assess the postural control on different floors with eyes open, eyes closed, and cognitive dual-task, ankle, and trunk proprioception, plantar sensation, and general cognitive status of patients diagnosed with Type 2 diabetes between the ages of 18-65, and to compare them with healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-65
* Volunteering to participate in researc
* Being diagnosed with Type 2 diabetes according to the criteria of the American Diabetes Association (ADA)

Exclusion Criteria:

* Insufficient cognitive level
* Traumatic nerve injury
* Presence of congenital anomaly in the upper extremity
* Presence of systematic disease (eg: rheumatological)
* Having a problem involving the neurological system
* Surgery involving the upper extremity in the last 6 months

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 31 patients between the ages of 18-65 who were diagnosed with Type 2 diabetes and 31 healthy participants who were not diagnosed with Type 2 diabetes, who applied to Hasan Kalyoncu University Application and Research Center, will participate in the study. All participants will be given detailed information about the study and signed a written informed consent form stating that they have voluntarily accepted the study.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2023-09-10 (Actual); Primary Completion 2023-11-10 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Postural Control | 20 minutes
  Postural control of the participants will be measured objectively by transferring the data taken from the body to the computer with the help of a wearable sensor using Gyko-Microgate software. Ellipsoid area and moving speed will be measured in mm² and mm/s².
Ankle proprioception | 10 minutes
  Proprioception in ankle plantar flexion and dorsiflexion will be measured with the help of a digital goniometer.
Lumbal proprioception | 5 minutes
  Proprioception in lumbar flexion and extension will be measured with the help of a digital goniometer.

SECONDARY OUTCOMES:
Plantar sensation | 5 minutes
  Semmes-Weinstein Monofilament Test
Cognitive status | 10 minutes
  Montreal Cognitive Assessment (MoCA) is evaluated out of 30 points. The highest score that can be obtained from the scale is 30, the lowest score is 0. 21 points is the reference limit and a value below 21 points indicates that there is an affect on cognitive status.
Dynamic Balance | 1 minute
  Timed Up and Go Test

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gorniak SL, Lu FY, Lee BC, Massman PJ, Wang J. Cognitive impairment and postural control deficit in adults with Type 2 diabetes. Diabetes Metab Res Rev. 2019 Feb;35(2):e3089. doi: 10.1002/dmrr.3089. Epub 2018 Nov 8. PMID 30338902